CLINICAL TRIAL: NCT05305703
Title: Effectiveness of Soft Tissue Mobilization and Trigger Point Release vs. Stretching on Tension-type Headache in University Students
Brief Title: Effectiveness of Soft Tissue Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Esha Khan, lecturer, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECCR/ Ref No.: BI-14/DPT2019
Record Dates: First submitted 2022-03-12; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical muscles Stretching (Experimental): Stretching is applied to the effected muscles in order to increase the muscle length and flexibility by breaking adhesions. Stretching exercises considerably decrease neck pain and improve range of motion
  Interventions: Other: cervical stretching
- Soft tissue mobilization with trigger point release. (Experimental): Soft tissue mobilization increases skin temperature, a rise in skin temperature indicates increase blood flow of involved area, provide relaxation and reduce muscle tension.Trigger point therapy is consisting of rubbing and pressing on trigger points.Heavy pressure must be applied to release trigger, light pressure is not effective. Pressure should be applied slowly and released slowly for best results and the pressure should be maintained until there is a change in pain
  Interventions: Other: soft tissue mobilization

INTERVENTIONS:
Other: cervical stretching — Heating therapy for 10 minutes Passive stretching of neck muscles including Sub-occipital muscles, Trapezius upper boarder and Sternocleidomastoid muscle with 10 reps each
  Arms: Cervical muscles Stretching
Other: soft tissue mobilization — Heating therapy for 10 minutes Soft tissue mobilization for 8 minutes and trigger point release of sub-occiptal muscles with 5 repetitions each.
  Arms: Soft tissue mobilization with trigger point release.

SUMMARY:
The aim of this study was to determine the effects of soft tissue mobilization and trigger point release verses stretching in tension-type headache among university students. Two randomized groups of participants with tension type headache will be treated with combination therapy of soft tissue mobilization and trigger point release therapy after the application of hot-pack in experimental group while control group received stretching of cervical muscles after hot-pack application .Both, male and female patients meeting the inclusion criteria will be included. Patients having malignancy and cervical tumor will be excluded.

DETAILED DESCRIPTION:
It was a Randomized Control Trial Study. Study setting was Bashir Institute of Health sciences. Inclusion Criteria was Age 18 to 25 year's students, with tension type headache and trigger point in neck muscles. 30 Subjects were randomly and equally allocated to experimental group (n=15) and control group (n=15) through toss and coin method. Outcomes include cervical range of motions were measured by Goniometer and VAS for paini.e., used at baseline and at the final session for duration of 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-25 years.
* Both Male and Female gender
* Trigger points in neck muscles

Exclusion Criteria:

* Patients taking pharmacologicaldrugs.
* Presence of co morbidities.
* Malignancy/ Trauma in cervical region
* Skin infections or open wound in cervical region

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
changes from baseline in Visual Analogue Scale | baseline and 3 weeks
  Reliability of Visual Analogue Scale for pain measurement

SECONDARY OUTCOMES:
changes from baseline in Goniometer | baseline and 3 weeks
  Goniometry is commonly used in clinical practice for assessment of range of motion and treatment interventions. It is used in patients who have insufficient range of motion due to muscletightness, joint stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Nasir khan, DPT, Principal Investigator — Bashir Institute of Health Sciences
Locations (1):
- Nasir khan, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No